CLINICAL TRIAL: NCT01315106
Title: High Resolution 3D Diffusion-weighted Breast MRI
Status: Terminated | Type: Observational
Why Stopped: Business Decision
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB-19595; SU-11152010-7211 (Other: Stanford University); BRS0013 (Other: OnCore); 5R21EB012591-02 (NIH)
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Magnetic Resonance Image Scanner — Magnetic Resonance Imaging; 1.5 Tesla or 3 Tesla MRI scanner
  Other Names: MRI

SUMMARY:
The purpose of this study is to determine how well a new MRI technique called "High resolution 3D diffusion-weighted breast MRI" detects breast cancer.

DETAILED DESCRIPTION:
The objective of this study is to assess the diagnostic accuracy of a new non-contrast MRI method for breast cancer detection. The study design is a single arm observational study. The new technique will be added on to the standard sequences that a women undergoes during a breast MRI. The resulting images will be compared with her standard breast MRI images, and with results of subsequent pathology.

ELIGIBILITY:
Inclusion Criteria:1. Patient scheduled for contrast-enhanced breast MRI to image possible breast cancer.

2. Female

3. Age >18 Exclusion Criteria:1. Lactation

2. Pregnancy

3. Patient undergoing chemotherapy. These patients are excluded because chemotherapy changes the biology of breast cancers. Since the ultimate objective of the research is to develop a new imaging method for breast MRI screening (detection of previously unknown tumors), results in treated tumors would not be relevant. Including treated tumors could yield a misleading assessment of the performance of the new method since treated tumors have different imaging characteristics than de novo tumors.

4. Patient scheduled for pre-operative chemotherapy. These patients are excluded if they are going to be treated only on the basis of fine needle aspiration. The project seeks to correlate all tumors detected with standard histopathology of their untreated neoplasm. This exclusion criteria will be very unusual because most patients planning neoadjuvant chemotherapy do so on the basis of a pre-chemo core needle biopsy, which provide adequate histopathologic proof necessary for enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stanford Radiology Department MRI facilities
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2014-01-07 (Actual); Study Completion 2014-01-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the new MRI method | 8 weeks
Lesion detection rate of the new MRI method | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruce L. Daniel, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States